CLINICAL TRIAL: NCT01604668
Title: Comparative Accuracy of Three Versions of Non-Invasive Hemoglobin Monitoring.
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 1000524C
Record Dates: First submitted 2012-05-18; First posted 2012-05-24 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RevF vs RevG vs Pronto-7: Comparison of hemoglobin levels derived by continuous hemoglobin sensor RevF versus continuous hemoglobin sensor RevG versus an intermittent hemoglobin level derived from the Pronto-7 hand-held device versus a hemoglobin derived from a blood sample.

SUMMARY:
There is no study hypothesis. The purpose of this study is to compare the accuracy of the: 1) SpHb (Radical 7 Pulse Co-Oximetry with SpHb™) RevF sensor (currently marketed), 2) the SpHb RevG sensor (a new, limited release version), and 3) the Pronto-7 sensor (currently marketed version) in patients undergoing spine surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare the accuracy of the: 1) SpHb RevF sensor (currently marketed), 2) the SpHb RevG sensor (a new, limited release version), and 3) the Pronto-7 sensor (currently marketed version) in patients undergoing spine surgery. The results from the three sensors will be compared to a blood hemoglobin level taken intermittently (as a function of the patient's anesthesia care) and analyzed in the UCSF Clinical Laboratories.

This is an observational study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ASA Classification 1, 2 or 3
* Scheduled to undergo spine surgery

Exclusion Criteria:

* Pregnant of nursing
* In the investigator's judgement would not be suitable for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison of hemoglobin levels derived by sensor RevF versus sensor RevG versus a hemoglobin derived from a blood sample. A baseline hemoglobin level will be taken from the Pronto-7 hand-held hemoglobin device prior to surgery. | Two or more measurements during surgery
  Comparison of hemoglobin levels derived by sensor RevF versus sensor RevG versus a hemoglobin derived from a blood sample. A baseline hemoglobin level will be taken from the Pronto-7 hand-held hemoglobin device prior to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D. Miller, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Moffitt/Long Hospitals, San Francisco, California, United States

REFERENCES:
- [Background] Miller RD, Ward TA, Shiboski SC, Cohen NH. A comparison of three methods of hemoglobin monitoring in patients undergoing spine surgery. Anesth Analg. 2011 Apr;112(4):858-63. doi: 10.1213/ANE.0b013e31820eecd1. Epub 2011 Mar 8. PMID 21385985